CLINICAL TRIAL: NCT04724681
Title: Continuous Wireless Monitoring of Vital Signs and Automated Alerts of Patient Deterioration in Patients Admitted With COVID-19 Infection
Acronym: WARD COVID-19
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of funding
Sponsor: University Hospital Bispebjerg and Frederiksberg (Other)
Collaborators: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Katja Kjær Grønbæk, Principal Investigator, University Hospital Bispebjerg and Frederiksberg
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H-20025357
Record Dates: First submitted 2020-10-21; First posted 2021-01-26 (Actual); Last update posted 2023-06-01 (Actual); Status verified 2023-05

CONDITIONS: Clinical Deterioration
MeSH Terms: conditions — Clinical Deterioration

STUDY DESIGN:
Intervention Model Description: A prospective controlled cohort study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Monitoring arm (Active Comparator): Patients in this arm will have their vital signs monitored with continuous wireless devices and patients in this arm will be monitored with standard Early Warning Score
  Interventions: Device: WARD CSS
- standard Early Warning Score arm (No Intervention): Patients in this arm will be monitored with standard Early Warning Score

INTERVENTIONS:
Device: WARD CSS — Wireless devices monitor vital signs continuously and transmit real-time data to an app that notifies clinical personnel when relevant deviations in vital signs occur This group will be monitored with standard Early Warning Score as well
  Arms: Monitoring arm

SUMMARY:
For patients admitted with COVID-19 infection, it is often difficult to predict if or when their clinical condition will deteriorate. However subtle changes in vital signs are usually present 8 to 24 hours before a life-threatening event such as respiratory failure leading to ICU admission, or unanticipated cardiac arrest. Such adverse trends in clinical observations can be missed, misinterpreted or not appreciated as urgent. New continuous and wearable 24/7 clinical vital parameter monitoring systems offer a unique possibility to identify clinical deterioration before patients condition progress beyond the point-of-no-return, where adverse events are inevitable. The primary aim of this study is to test the effect of continuous wireless vital signs monitoring with generation of real-time alerts through a purpose-built GUI, compared to standard EWS monitoring on the cumulative duration of any severely deviating vital signs

ELIGIBILITY:
Inclusion criteria

* Adult patients (≥18 years).
* Inclusion possible within 72 hours of admission, OR within 48 hours of discharge from an ICU to a medical ward
* At least one expected overnight stay.
* Patient admitted with confirmed COVID-19 infection

Exclusion criteria

* Patient expected not to cooperate with study procedures.
* Allergy to plaster or silicone.
* Patients admitted for palliative care only (i.e. no active treatment).
* Patients previously enrolled in the studies WARD-COPD (H-18026653) or WARD-Surgery (H-17033535).
* Inability to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2020-11-03 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Cumulative duration of deviating vital signs: SpO2 < 85% min-1 | up to 16 days
  Cumulative duration in minutes of the following deviations in vital signs during the monitoring period:
  ● SpO2 < 85% min-1
Cumulative duration of deviating vital signs, respiratory rate ≤ 5 min-1 | up to 16 days
  Cumulative duration in minutes of the following deviations in vital signs during the monitoring period:
  ● Respiratory rate ≤ 5 min-1
Cumulative duration of deviating vital signs, respiratory rate > 24 min-1 | up to 16 days
  Cumulative duration in minutes of the following deviations in vital signs during the monitoring period:
  ● Respiratory rate > 24 min-1
Cumulative duration of deviating vital signs, heart rate > 130 min-1 | up to 16 days
  Cumulative duration in minutes of the following deviations in vital signs during the monitoring period:
  ● Heart rate > 130 min-1
Cumulative duration of deviating vital signs, heart rate ≤ 30 min-1 | up to 16 days
  Cumulative duration in minutes of the following deviations in vital signs during the monitoring period:
  ● Heart rate ≤ 30 min-1
Cumulative duration of deviating vital signs, ScO2 | up to 16 days
  Cumulative duration in minutes of the following deviations in vital signs during the monitoring period:
  ● Lowest ScO2 (mean for ≥ 5 mins) min-1

SECONDARY OUTCOMES:
Frequency of predefined microevents (deviating vital signs) | up to 16 days
  The frequency of micro events (deviating vital signs), measured by continuous vital sign monitoring and as measured by EWS in the control group
  The microevents are defined as follows, and the the outcome are frequency of these
  * RR ≤5 bpm AND HR >20 bpm
  * RR ≥24 bpm
  * RR <11 bpm AND SpO2 <88 %
  * SpO2 <80%
  * SpO2 <85%
  * SpO2 <88%
  * SpO2 <92%
  * HR >130 bpm
  * HR ≥111 bpm
  * HR <30 bpm
  * HR = 30-40 bpm
  * Atrialflutter
Change in vital parameters | up to 16 days
  Change in vital parameters one hour following an alarm as defined below
  Desaturation
  • Change in SpO2 60 minutes after an alarm has been triggered. (SpO2 < 85 % for more than 5 minutes, SpO2 < 80 % for more than 1 minutes, SpO2 < 88 % for more than 10 minutes )
  Tachypnea
  • Change in RR 60 minutes after an alarm has been triggered. (RR >24 bpm for more than 5 minutes)
  Bradypnea/apnea • Change in RR and HR 60 minutes after an alarm has been triggered (RR ≤5 bpm AND HR >20 bpm for more than one minute)
  Hypoventilation • Change in RR and SpO2 60 minutes after an alarm has been triggered. (RR <11 bpm AND SpO2 <88% for more than 5 minutes )
  Tachycardia
  • Change in HR 60 minutes after an alarm has been triggered. (HR >130 for more than 30 minutes, HR >111 for more than 60 minutes)
  Bradycardia
  • Change in HR 60 minutes after an alarm has been triggered. (HR <30 bpm for more than 1 minutes, HR 30-40 bpm for more than 5 minutes)
The frequency of events with desaturation as defined below and the simultaneous values of ScO2 | up to 16 days
  The frequency of events with desaturation as defined below and the simultaneous values of ScO2
  * SpO2 <80% >1 min
  * SpO2 <85% > 5 min
  * SpO2 <88% > 10 min
  * SpO2 <92% > 60 min
Events with ScO2 < 60% for ≥ 1 min | up to 16 days
  The frequency of events with ScO2 < 60% for ≥ 1 min and the simultaneous measured SpO2 values

OTHER OUTCOMES:
Duration of vital sign deviation | up to 16 days
  Duration of each of the following vital sign deviations
  * SpO2 < 85%
  * Respiratory rate ≤ 5 min-1
  * Respiratory rate > 24 min-1
  * Heart rate > 130 min-1
  * Heart rate ≤ 30 min-1
  * Lowest ScO2 (mean for ≥ 5 mins)
ECG pattern after alarm | up to 16 days
  ECG pattern one hour following an AFLI alarm. (analysed with paired statistics within the continuously monitored group). The ECG pattern one hour following an alarm can be classified as either normal sinusrythm or AFLI
Adverse clinical ooutcomes | 6 months
  Any adverse clinical outcomes as defined in the protocol
Response to an alarm | up to 16 days
  Staff response time to an alarm (stratified according to time of day)
Contact to the attending doctor on call | up to 16 days
  number of times that the attending doctor on call is contacted during admission
Contact to intensive care physician on call | up to 16 days
  number of times that the intensive care physician on call is contacted during admission
Activation of Emergency Response Team | up to 16 days
  number of times that the Emergency Response Teams is activated during admission
Invasive ventilation | up to 16 days
  The frequency of invasive ventilation during admission
ICU admissions | up to 16 days
  The frequency of ICU admissions during admission
Length of stay | up to 16 days
  Length of stay (LOS) in days
Cumulative duration of ScO2 <60 % during admission | up to 16 days
  Cumulative duration of ScO2 < 60 % related to the total time of NIRS monitoring

CONTACTS AND LOCATIONS:
Overall Officials: Katja Grønbæk, MD, PhD-student, Principal Investigator — Bispebjerg Hospital
Locations (1):
- Bispebjerg and Frederiksberg Hospital, Copenhagen, Denmark